CLINICAL TRIAL: NCT03641859
Title: Evaluation of Pain and Anxiety in Patients With an Invasive Procedure in Emergencies: Randomized Trial
Brief Title: Evaluation of Pain and Anxiety in Patients With an Invasive Procedure in Emergencies
Acronym: URGENCES_RV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URGENCES_RV
Record Dates: First submitted 2018-08-13; First posted 2018-08-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Virtual Reality
Keywords: pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthesia (No Intervention): The study population will consist of consecutive pre-screened patients when they arrive at the emergency department at the level of the host nurse. The emergency physician who will be in charge of the patient gives the patient the information form and ensures the absence of contraindication, responds to the patient's questions and collects his free, informed and express consent.
  Once the patient is included, the group (with or without virtual reality) of the patient's participation in the study will be notified by the reception nurse and emergency referral:
  - Arm 1 (usual care): the procedure of care will be the same as usual.
- local anesthesia + virtual reality (Experimental): The study population will consist of consecutive pre-screened patients when they arrive at the emergency department at the level of the host nurse. The emergency physician who will be in charge of the patient gives the patient the information form and ensures the absence of contraindication, responds to the patient's questions and collects his free, informed and express consent.
  Once the patient is included, the group (with or without virtual reality) of the patient's participation in the study will be notified by the reception nurse and emergency referral:
  - Arm 2 (intervention): local anesthesia + virtual reality
  Interventions: Device: virtual reality

INTERVENTIONS:
Device: virtual reality — The virtual reality headset can be used for 45 minutes with the need to pause for 5 minutes if the gesture lasts longer. The VR sequence will be complete when the end of the programmed time is reached to preserve the patient's immersion. The patient will be able to see the final sequence at the end of the gesture in order to get used to the real world again. The programs and their durations will be adjusted to the duration of the gesture concerned. Regarding the pain, anxiety and satisfaction visual analogue scales, they will be performed just after the removal of the VR helmet.
  Virtual reality videos are from Healthy Mind® software. The videos are contemplative with three kinds of relaxing landscapes accompanied by a sound universe specifically composed to relax the patient. The patient can choose one of three interactive worlds (an Asian garden, a forest or a mountain).
  Arms: local anesthesia + virtual reality

SUMMARY:
A large number of patients presenting to the emergency department will have an invasive or potentially painful treatment (suture, urinary catheterization, reduction of dislocation or fracture). This care is a source of pain and anxiety for patients.

Since 1998, the management of pain is a public health priority in France. Law No. 2002-3003 of 4 March 2002 on the rights of the sick and the quality of the health system has made pain management a right: "Everyone has the right to receive care to relieve his pain. This must be in all circumstances prevented, evaluated, taken into account and treated ".

In emergency departments, the use of antalgic drug treatments and local anesthetics is systematic.

DETAILED DESCRIPTION:
Other techniques to create diversions proposed in the recommendations of the French Society of Emergency Medicine for the management of wounds in emergencies can be used to improve the experience of patients: the use speech during the gesture or certain forms of hypnosis.

Pain and anxiety are two important factors to integrate to improve the management of patients in emergencies.

To improve pain and anxiety, distraction is a technique that can be used. Virtual reality is a distraction technique not yet frequently used but studied. It combines the visual and the auditory allowing immersion in a virtual world thanks to a helmet retranscribing a three-dimensional image. The diversion of attention through the use of virtual reality allows the patient to immerse themselves in a fictional environment through a mask on the eyes inhibiting the vision of the outside world and a headphone reducing external sounds and reinforcing the mechanism of 'immersion.

The use of the virtual reality headset has already shown benefits during pain care in burn patients and children.

The virtual reality headset has not yet been studied as a distraction tool for invasive and potentially painful care in emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman (age ≥ 18 years)
* Francophone
* Patient with medical insurance
* Patient with a wound requiring trunk or limb sutures
* Or male patient requiring an urinary catheter
* Patient with cutaneous and subcutaneous wounds (deep plane possible) but without repair of noble tissues (tendons or fasciae) with no limit on the number of points to be made (i.e. without impact on the main endpoint).

Exclusion Criteria:

* Patient with a wound or skin infection of the face
* Patients with nausea, vomiting, dizziness
* Patients with a history of neurological disorders with epilepsy
* Patient whose investigator judges that he can not wear a virtual reality helmet
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Analogical visual scale on the pain felt during the treatment | 1 hour after the beginning of virtual reality
  Analogical visual scale on the pain felt during the treatment Analogical Visual Scale (EVA): a slider that allows the patient to self-assess the pain felt by a slider On the front of the ruler, is drawn a line or a pyramid on which the patient moves the cursor from the end "no pain" to the end "maximum pain imaginable" On the back of the slide, the caregiver reads the pain felt by the patient using a graduation in millimeters (from 0 to 100 mm)

SECONDARY OUTCOMES:
Analogical visual scale evaluating the patient's anxiety during the treatment | 1 hour after the beginning of virtual reality
  Analogical visual scale evaluating the patient's anxiety during the treatment Analogical Visual Scale (EVA): a slider that allows the patient to self-assess the anxiety felt by a slider On the front of the ruler, is drawn a line or a pyramid on which the patient moves the cursor from the end "no anxiety" to the end "maximum anxiety" On the back of the slide, the caregiver reads the pain felt by the patient using a graduation in millimeters (from 0 to 100 mm)
Analogical visual scale of patient satisfaction and satisfaction questionnaire | 1 hour after the beginning of virtual reality
  Analogical visual scale of patient satisfaction and satisfaction questionnaire Analogical Visual Scale (EVA): a slider that allows the patient to self-assess the pain felt by a slider On the front of the ruler, is drawn a line or a pyramid on which the patient moves the cursor from the end "not satisfied" to the end "very satisfied" On the back of the slide, the caregiver reads the pain felt by the patient using a graduation in millimeters (from 0 to 100 mm)
Analogical visual scale evaluating anxiety and pain before and after the gesture according to the treatment group | 1 hour after the beginning of virtual reality and 1 hour before the end of virtual relaity
  Analogical visual scale evaluating anxiety and pain before and after the gesture according to the treatment group Analogical Visual Scale (EVA): a slider that allows the patient to self-assess the pain felt by a slider On the front of the ruler, is drawn a line or a pyramid on which the patient moves the cursor from the end "no pain/anxiety" to the end "maximum pain imaginable/maximum anxiety" On the back of the slide, the caregiver reads the pain felt by the patient using a graduation in millimeters (from 0 to 100 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie MARTEAU, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Uman LS, Birnie KA, Noel M, Parker JA, Chambers CT, McGrath PJ, Kisely SR. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD005179. doi: 10.1002/14651858.CD005179.pub3. PMID 24108531
- [Result] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Result] Hoffman HG, Patterson DR, Soltani M, Teeley A, Miller W, Sharar SR. Virtual reality pain control during physical therapy range of motion exercises for a patient with multiple blunt force trauma injuries. Cyberpsychol Behav. 2009 Feb;12(1):47-9. doi: 10.1089/cpb.2008.0056. PMID 19018695
- [Result] Schneider SM, Workman ML. Virtual reality as a distraction intervention for older children receiving chemotherapy. Pediatr Nurs. 2000 Nov-Dec;26(6):593-7. PMID 12026359
- [Result] Miller KM, Wysocki T, Cassady JF Jr, Cancel D, Izenberg N. Validation of measures of parents' preoperative anxiety and anesthesia knowledge. Anesth Analg. 1999 Feb;88(2):251-7. doi: 10.1097/00000539-199902000-00005. PMID 9972736
- [Result] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420